CLINICAL TRIAL: NCT05305495
Title: Empagliflozin for Patients With Acutely Decompensated Congestive Heart Failure, Diuretic Resistance, and Moderate to Advanced Chronic Kidney Disease
Brief Title: Empagliflozin in Acute Heart Failure
Acronym: DRIP-AHF-1
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Thomas Mavrakanas, Assistant Professor, Junior Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-8411
Record Dates: First submitted 2022-03-04; First posted 2022-03-31 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Acute Heart Failure; Chronic Kidney Diseases
Keywords: Empagliflozin; Acute Heart Failure; Chronic kidney disease; Diuretic resistance; Furosemide
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, single arm, cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with diuretic resistance (Experimental)
  Interventions: Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Patients who fulfill the inclusion criteria will receive an intravenous dose of 1.0-1.5 mg/kg of furosemide (≤120 mg) and urine output will be monitored for three hours. Those with a urine output < 300 ml in the first two hours post furosemide administration will receive a single oral dose of 25 mg of empagliflozin. Two hours after taking empagliflozin, patients will receive a second intravenous dose of 1.0-1.5 mg/kg of furosemide with another timed urine collection at three hours. Empagliflozin will then be continued daily for five days or until hospital discharge, unless the treating physician considers this not to be clinically appropriate.
  Other Names: Jardiance (DIN: 02443945)

SUMMARY:
The objective is to study in a prospective, interventional, single arm, cohort study the potential synergistic diuretic effect of empagliflozin, in addition to furosemide, in hypervolemic patients admitted with acutely decompensated heart failure and diuretic resistance at the McGill University Health Centre (MUHC).

The investigators hypothesize that the sodium-glucose cotransporter-2 (SGLT-2) inhibitor empagliflozin will enhance the diuretic effect of furosemide in patients with acutely decompensated heart failure, moderate to advanced chronic kidney disease, and underlying diuretic resistance, as identified by the three-hour urine output post diuretic administration on the first day of the study, compared with furosemide alone.

ELIGIBILITY:
Inclusion Criteria (all have to apply) :

* moderate to advanced CKD, defined as an eGFR <45 ml/min/1.73m2; The average creatinine values over the last 12 months will be used to calculate baseline eGFR.
* acutely decompensated heart failure, defined as dyspnea at rest or with minimal physical activity, associated with at least one clinical sign of congestion and at least one objective measure of heart failure (pulmonary-capillary wedge pressure >20 mm Hg or evidence of pulmonary congestion on chest radiography or brain natriuretic peptide (BNP) level ≥400 pg/ml or N-terminal pro-BNP level ≥1000 pg/ml);
* evidence of inadequate response to loop diuretics, defined as a urine output < 1000 ml/24h or a weight loss < 1kg /24h. For patients who have not received loop diuretics, a furosemide stress test can be conducted.
* stable hemodynamics, defined as systolic blood pressure >90 mmHg and/or mean arterial pressure >65 mmHg in the absence of intravenous norepinephrine or epinephrine in the last 24 hours.

Exclusion Criteria:

* new use of a non-loop diuretic other than an MRA
* history of type 1 diabetes mellitus
* euglycemic diabetic ketoacidosis
* liver disease defined by serum levels of transaminases or alkaline phosphatase more than three times the upper limit of normal at screening
* known hypersensitivity to SGLT-2 inhibitors
* use within the last 48 h of an SGLT-2 inhibitor or a combined SGLT-1 and SGLT-2 inhibitor
* maintenance dialysis or need for emergent renal replacement therapy
* gastrointestinal surgery or gastrointestinal disorder that could interfere with trial medication absorption
* recurrent severe genital or urinary tract infection
* pregnancy or breastfeeding
* any other clinical condition that would jeopardize patient safety while participating in this trial
* Patients with an acute rise in creatinine levels (acute cardiorenal syndrome) upon presentation will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Diuretic effect of empagliflozin in association with furosemide | Day 1
  Three-hour urine output post empagliflozin-furosemide administration, compared with furosemide alone

SECONDARY OUTCOMES:
Fractional excretion of sodium in the urine | Day 1
  FeNa (%)
Total urine sodium output | Day 1-5
  Urine sodium per 24h
Changes in volume status | Day 1-5
  Net fluid balance
Incidence of AKI | Day 1-5
  Using the conventional KDIGO criteria
Electrolyte abnormalities - Sodium | Day 1-5
  Concentration of sodium
Electrolyte abnormalities - Potassium | Day 1-5
  Concentration of potassium
Electrolyte abnormalities - Magnesium | Day 1-5
  Concentration of magnesium

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mavrakanas, MD, Principal Investigator — Research Institute of the McGill University Health Center
Locations (1):
- Research Institute of the McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No